CLINICAL TRIAL: NCT05152615
Title: A Pilot Proof of Concept Study of the Effects of Administration of a Short Chain Fatty Acid (SCFA) in Rheumatoid Arthritis (EASi-RA)
Brief Title: A Pilot Proof of Concept Study of the Effects of Administration of SCFA in Rheumatoid Arthritis (EASi-RA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-02068
Record Dates: First submitted 2021-12-01; First posted 2021-12-10 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Short Chain Fatty Acid (SCFA); Butyrate; Gut Microbiome
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Fatty Acids, Volatile; Dietary Supplements; Butyrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- New Onset Rheumatoid Arthritis (NORA) Patient (Experimental): NORA patients receiving methotraxate as first line therapy (standard of care) will take additional oral SCFA supplementation for the purposes of the study.
  Interventions: Dietary Supplement: Short Chain Fatty Acids (SCFA) Dietary Supplement

INTERVENTIONS:
Dietary Supplement: Short Chain Fatty Acids (SCFA) Dietary Supplement — Butryate 1000 mg three times daily will be used in this study.
  Other Names: Butyrate

SUMMARY:
This study is a pilot, proof of concept study to determine the effects of administering an oral short chain fatty acid (SCFA) supplement along with methotrexate as first line treatment of new onset rheumatoid arthritis (NORA) patients. Up to 50 participants will be included to obtain a sample size of at least 16 participants taking the oral supplement. The study team hypothesizes that oral SCFA will change the participants' gut microbiome and regulatory immune responses. Clinical data to assess for adverse events, stool, urine samples and peripheral blood will be collected at baseline, 2 and 4 months with an optional 6-month time point. Fecal microbiome will be analyzed. Adaptive immune responses will be analyzed from participant blood samples.

ELIGIBILITY:
Inclusion Criteria:

1. New diagnosis of rheumatoid arthritis (RA) (<6 months) meeting 2010 ACR/EULAR for RA
2. Scheduled to begin treatment with methotrexate at any dose as standard medical care
3. Able and willing to provide written informed consent prior to any study specific procedures
4. Age 18 years and above at time of enrollment
5. Subjects not excluded based on race or ethnicity

Exclusion Criteria:

1. Participants who are pregnant or are currently breastfeeding
2. History of sensitivity to study compound or any of their excipients
3. Previous intolerance to SCFA or related compounds
4. Current (within 3 months of screening) treatment with csDMARDs
5. Current or past (ever) treatment with biologic therapies (including but not limited to anti-TNF, anti-IL-17, anti-IL-12/23)
6. Current antibiotic treatment (within 3 months of screening)
7. Current consumption of probiotics (within 3 months of screening)
8. Severe hepatic impairment (eg, ascites and/or clinical signs of coagulopathy)
9. Renal failure (eGFR <30 or requiring dialysis) by history
10. History of other autoimmune disease
11. Current immunodeficiency state (e.g., cancer, HIV, others)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Change in Percentage of Circulating T Regulatory Cells (Treg) | Baseline, Visit 2 (60 days)

SECONDARY OUTCOMES:
Change in gut microbiota composition after SCFA supplementation | Baseline, Visit 2 (60 days), Visit 3 (120 days), Visit 4 (180 days)
Change in Fecal SCFA Concentration after SCFA supplementation | Baseline, Visit 2 (60 days), Visit 3 (120 days), Visit 4 (180 days)
Change in Interleukin-10 (IL-10) Production Levels after SCFA Supplementation | Baseline, Visit 2 (60 days), Visit 3 (120 days), Visit 4 (180 days)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Scher, MD, Principal Investigator — NYU Langone Health; Rebecca B Blank, MD, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be available upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to Rebecca.Blank@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.